CLINICAL TRIAL: NCT02229656
Title: Olaparib Dose Escalation Trial in Patients Treated With Radiotherapy for Stage II-III Laryngeal and Stage II-III HPV-negative Oropharyngeal Squamous Cell Carcinoma
Brief Title: Olaparib and Radiotherapy in Head and Neck Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N13ORH; 2011-002963-79 (EudraCT Number)
Record Dates: First submitted 2014-08-28; First posted 2014-09-01 (Estimated); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Laryngeal Cancer Stage II; Laryngeal Cancer Stage III; Carcinoma, Squamous Cell; Head and Neck Neoplasms
Keywords: olaparib; radiotherapy; Laryngeal SCC; oropharyngeal SCC
MeSH Terms: conditions — Laryngeal Neoplasms; Carcinoma, Squamous Cell; Head and Neck Neoplasms | interventions — Radiotherapy; olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- radiotherapy and olaparib (Experimental): Radiotherapy will be given with accelerated fractionation following the DAHANCA schedule Olaparib: dose escalation
  Interventions: Radiation: radiotherapy; Drug: Olaparib

INTERVENTIONS:
Radiation: radiotherapy — Primary tumor and lymph nodes will receive 35 fractions of 2 Gy resulting in a total dose of 70 Gy. Elective fields will receive 35 fractions of 1.55 Gy resulting in a total dose of 54.25 Gy in case a SIB technique is used, or 23 fractions of 2 Gy resulting in a total dose of 46 Gy in case a sequential boost technique is used. The higher total prescribed physical dose to the elective fields in a SIB technique based RT plan compensates for the lower dose per fraction and results in an equal biological effective dose when compared with a sequential boost technique.
Drug: Olaparib — The pre-defined dose levels of olaparib are 25mg QD, 25, 50, 100, 200, and 300 mg BID
  Other Names: AZD2281; KU-0059436

SUMMARY:
Accelerated, normofractionated radiotherapy is the treatment of choice in stage II-III laryngeal and oropharyngeal squamous cell carcinoma (SCC). However, twenty to thirty percent of patients with stage II-III laryngeal and HPV negative oropharyngeal SCC develop disease progression, mainly due to lack of locoregional control. Radiosensitizers such as cisplatin and cetuximab are added to radiotherapy in more advanced stage of head and neck (H&N) cancer. These radiosensitizers improve loco-regional control and overall survival. Unfortunately, as these radiosensitizers, notably cisplatin, also dose intensify the radiation dose in normal tissues, they also significantly increase toxicity. Adding a more tumor-specific radiosensitizing agent could improve loco-regional control and overall survival without significantly increasing toxicity.

Radiotherapy kills tumor cells by inducing DNA damage. The efficacy of radiotherapy is limited by the ability of tumor cells to repair this DNA damage. Poly(ADP-ribose)polymerase (PARP) is an essential enzyme in base excision repair and single strand break DNA repair, DNA lesions arising from radiation treatment. PARP inhibition and consequently the inhibition of PARP-facilitated DNA repair enhances the anti-tumor activity of radiotherapy, as shown in preclinical studies including head and neck xenograft studies. This radiosensitization is thought to be proliferation dependent and is more pronounced in homologous recombination (HR) deficient cells, providing an opportunity for tumor specific targeting. Genetic analyses suggest that HR deficiency is commonly found in H&N SCC: ATM loss has been reported in 60% of human H&N SCC biopsies and FANC-F defects were reported in 15-21% of human H&N SCC biopsies and cell lines.

The efficacy of radiotherapy is also limited by tumor hypoxia, as tumor hypoxia results in radioresistance. Some PARP inhibiting compounds increase tumor perfusion in xenograft models, thereby reducing hypoxia and specifically sensitizing tumor cells to radiotherapy. Hypoxia is commonly found in H&N SCC and a high pre-treatment hypoxic fraction in H&N SCC tumors is associated with worse outcome. The high prevalence of both hypoxia and HR deficiencies in H&N SCC support the concept of tumor-specific radiosensitization by PARP inhibition in head and neck cancer patients.

Olaparib is a potent PARP inhibitor developed as an anti-cancer drug for HR defected tumors and as a dose intensifier for chemo- and radiotherapy. In humans, olaparib has a low toxicity profile as a single agent, with increasing bone marrow toxicity when combined with chemotherapy. The combination of olaparib and radiotherapy for H&N SCC is expected to improve locoregional control and thereby overall survival. However, this combination treatment has never been tested in humans before. The purpose of this study is to determine the safety and tolerability of radiotherapy for stage II-III laryngeal and stage II-III HPV-negative oropharyngeal SCC with concurrent olaparib.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Histologically confirmed squamous cell carcinoma of the larynx stage II-III (T2N0M0 or T1-2N1M0 or T3N0-1M0) or histologically confirmed squamous cell carcinoma of the oropharynx stage II-III (T1-2N1M0 or T3N0-1M0)
* In case of oropharyngeal carcinoma: tumor HPV status negative
* WHO performance 0-1
* Life expectancy of at least 6 months
* Adequate hematological, renal and hepatic functions

  * Hemoglobin ≥ 6.2 mmol/l
  * Leucocytes 3.0 x 10E9/l
  * Absolute neutrophil count 1.5x10E9/l
  * Platelet count 100 x 10E9/l
  * Total bilirubin ≤ 1.5 x UNL
  * ASAT/ALAT ≤ 2.5 x UNL
  * Creatinine clearance 50 ml/min; measured using a 24-hours urine sample or calculated using the Cockcroft-Gault formula
* Evidence of non-childbearing status for women of childbearing potential: negative urine or serum pregnancy test within 21 days of study treatment. Non-childbearing potential or postmenopausal is defined as:

  * Amenorrheic for 1 year or more following cessation of exogenous hormonal treatments
  * LH and FSH levels in post menopausal range for women under 50 years of age
  * Radiation-induced oophorectomy with last menses > 1 year ago
  * Chemotherapy-induced menopause with > 1 year interval since last menses
  * Surgical sterilisation (bilateral oophorectomy or hysterectomy)
* Patients of reproductive potential must agree to practice two effective medically approved contraceptive method during the trial and 3 months afterwards
* Signed written informed consent.

Exclusion Criteria:

* Patients eligible for concurrent chemoradiotherapy rather than radiotherapy alone
* Concurrent active malignancy other than localized, non-melanoma skin cancer or carcinoma-in-situ of the cervix (unless definitive treatment was completed 3 years or more before study entry and the patient has remained disease free)
* Anti-cancer therapy including chemotherapy, radiotherapy, endocrine therapy, immunotherapy or use of other investigational agents within the 3 weeks prior to start of therapy (or a longer period depending on the defined characteristics of the agents used e.g. 6 weeks for mitomycin or nitrosourea). Patients may continue the use of LHRH agonists for cancer; bisphosphonates for bone disease and corticosteroids.
* Major surgery within two weeks of starting study treatment.
* Participation in other trial with investigational drug or treatment modality
* Gastrointestinal disorders that may interfere with absorption of the study drug or patients who are not able to take oral medication.
* Tube feeding before the start of treatment.
* Prior radiotherapy to head & neck region.
* Blood transfusion in the four weeks prior to study entry
* Persistent toxicities (CTC ≥ grade 2) with the exception of alopecia, caused by previous cancer therapy
* QT-interval >470 msec
* Significant cardiovascular disease as defined by:

  * History of congestive heart failure defined as NYHA class III
  * History of unstable angina pectoris or myocardial infarction up to 3 months prior to trial entry;
  * Presence of severe valvular heart disease
  * Presence of a ventricular arrhythmia requiring treatment;
  * Uncontrolled hypertension
* Patients considered a poor medical risk due to:

  * non-malignant systemic disease
  * active, uncontrolled infection requiring parenteral antibiotics
  * a serious, uncontrolled medical disorder; examples include, but are not limited to:

    * uncontrolled major seizure disorder
    * unstable spinal cord compression
    * superior vena cava syndrome
    * extensive bilateral lung disease on HRCT scan
    * any psychiatric disorder that prohibits obtaining informed consent.
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.
* Patients who are known to be serologically positive for human immunodeficiency virus (HIV) and are receiving antiviral therapy.
* Patients with known active hepatic disease (i.e. Hepatitis B or C)
* Patients with myelodysplastic syndrome/acute myeloid leukaemia or features suggestive of MDS/AML on peripheral blood smear.
* Concomitant medications:

  * Any previous treatment with a PARP inhibitor, including olaparib
  * Patients receiving the following classes of inhibitors of CYP3A4 (see paragraph 6.4.2 for guidelines and wash out periods)

    * Azole antifungals
    * Macrolide antibiotics
    * Protease inhibitors
* Breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-09-24 (Actual); Primary Completion 2020-01-14 (Actual); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of dose limiting toxicities | 1 year
  * Blood transfusion dependency as judged by the PI, unless the patient has progressive disease
  * Development of MDS/AML
  * Grade ≥ 4 dysphagia
  * Grade ≥ 3 hemorrhage, aspiration, skin atrophy, trismus, osteoradionecrosis, radiation dermatitis, pneumonitis
  * Grade ≥ 2 fistula, myelitis
  * Grade ≥ 2 mucosal ulcer present ≥ 6 months after end of treatment
  * Fibrosis limiting joint or orifice movement (e.g. mouth) and/or limiting self care ADL
  * Only in patients with oropharynx SCC: grade ≥ 3 larynx stenosis
  * Any other (non-)hematological toxicity, which in the judgment of the Investigator is viewed as DLT; excluding fatigue

SECONDARY OUTCOMES:
acute toxicity | until 3 months after treatment
  severity, duration and relation with treatment of all adverse events according to CTCAE version 4.03
late toxicity | 3 months until 2 year after treatment
  severity, duration and relation with treatment of possibly, probably or definitely related adverse events according to CTCAE version 4.03

CONTACTS AND LOCATIONS:
Overall Officials: Marcel Verheij, MD, PhD, Principal Investigator — The Netherlands Cancer Institute
Locations (1):
- The Netherlands Cancer Institute, Amsterdam, Netherlands

REFERENCES:
- [Derived] de Haan R, van Werkhoven E, van den Heuvel MM, Peulen HMU, Sonke GS, Elkhuizen P, van den Brekel MWM, Tesselaar MET, Vens C, Schellens JHM, van Triest B, Verheij M. Study protocols of three parallel phase 1 trials combining radical radiotherapy with the PARP inhibitor olaparib. BMC Cancer. 2019 Sep 10;19(1):901. doi: 10.1186/s12885-019-6121-3. PMID 31500595